CLINICAL TRIAL: NCT05125640
Title: Randomized, Two-Sequence, Two-Treatment, Four-Period, Open-Label, Single Oral Dose, Crossover Bioequivalence Study of Progesterone 200 mg Soft Capsule vs Utrogestan® in Healthy Female Subjects Under Fasting Conditions
Brief Title: Fasting Bioequivalence Study of 2 Oral Progesterone Soft Capsules 200 mg in 48 Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joint Stock Company "Farmak" (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FK/BE/PROG/19
Record Dates: First submitted 2021-11-08; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Pharmacokinetics
Keywords: bioequivalence; pharmacokinetics; generic drugs; Progesterone; Soft Capsule; oral dosage form
MeSH Terms: interventions — Progesterone; Utrogestan

STUDY DESIGN:
Intervention Model Description: Comparative, Randomized, Two-Sequence, Two-Treatment, Four-Period, Open-Label, Single oral Dose, Fully Replicated, Crossover bioequivalence Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Progesterone 200 mg Soft Capsule (JSC "Farmak", Ukraine)
  Interventions: Drug: Progesterone 200 mg Soft Capsule (JSC "Farmak", Ukraine)
- Treatment B (Active Comparator): Utrogestan® 200 mg Soft Capsule (Manufacturer by: Cyndea Pharma, S.L., Spain, MAH: Laboratoires Besins International, France)
  Interventions: Drug: Utrogestan® 200 mg Soft Capsule (Manufacturer by: Cyndea Pharma, S.L., Spain, MAH: Laboratoires Besins International, France)

INTERVENTIONS:
Drug: Progesterone 200 mg Soft Capsule (JSC "Farmak", Ukraine) — Orally, with 240 mL of water at dosing in sitting position
  Other Names: Injesta
  Arms: Treatment A
Drug: Utrogestan® 200 mg Soft Capsule (Manufacturer by: Cyndea Pharma, S.L., Spain, MAH: Laboratoires Besins International, France) — Orally, with 240 mL of water at dosing in sitting position
  Other Names: Utrogestan®
  Arms: Treatment B

SUMMARY:
This study was designed to assess the bioequivalence of single oral dose of Progesterone 200 mg Soft Capsule (JSC "Farmak", Ukraine) Versus Utrogestan® 200 mg Soft Capsule (Manufacturer by: Cyndea Pharma, S.L., Spain, MAH: Laboratoires Besins International, France) In healthy female subjects under fasting conditions

DETAILED DESCRIPTION:
An open-label, randomized, single dose, two-treatment, four-period, two-sequence, fully replicated crossover bioequivalence study with a washout period of 7 days in healthy postmenopausal female subjects under fasting conditions.

During each period 26 blood samples were drawn 5 mL at (-1.00, -0.50, -0.137) before dosing and at 0.50, 1.00, 1.50, 2.00, 2.33, 2.67, 3.00, 3.50, 4.00, 4.50, 5.00, 5.50, 6.00, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 24.00, 48.00, 72.00 and 96.00 hours after dosing.

Mode of administration: Orally, with 240 mL of water at dosing in sitting position

Bioequivalence Acceptance Criteria:

▲Cmax (Maximum plasma concentration): Scaled average bioequivalence will be performed. Bioequivalence limits will be defined and widened according to the variance of σw2 within subject variability for the reference based on corrected progesterone.

AUC0-last (the area under the plasma concentration-time curve): The 90% confidence interval for this measure lies within an acceptance range of 80.00% - 125.00% based on corrected Progesterone.

▲Based on Cmax CVR% (Coefficient of Variation Ratio )=50.97% the calculated confidence interval acceptance limits were (69.83%-143.19%)

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers or past-smokers (an ex-smoker is defined as someone who has completely stopped using nicotine products, including nicotine cessation therapy, for at least 180 days prior to the first study drug administration).
* Body mass index (BMI) between 18.5 and 30 kg/m2 inclusive, and body weight not less than 45 kg (on the day of screening).
* Subject is available for the whole study and has provided her written informed consent.
* Subject is in good health as determined by screening medical history, physical examination, vital signs assessment (pulse rate, systolic and diastolic blood pressure and body temperature) and 12-lead ECG.Minor deviations outside the reference ranges will be acceptable, if dement not clinically significant by the Investigator.
* Acceptance of use of contraceptive measures during the whole study.
* Caucasian race.
* Normal liver and kidney functions tests. (On Screening).
* Results of laboratory tests (Prothrombin time (PT) and activated partial thromboplastin time (APTT), Thrombin Time (TT) tests also Erythrocyte sedimentation rate (ESR) and Hormones (follicle-stimulating hormone (FSH), luteinizing hormone (LH), Estradiol, Progesterone and Prolactin hormone (PRL)) results are within normal range or being assessed as clinically non-significant by the attending physician.(On Screening)

Exclusion Criteria:

* Known cardiovascular disease or history of hypotension.
* History of gout, urolithiasis, nephrolithiasis and hyperuricemia.
* Gastrointestinal diseases including gastric ulcer, renal or hepatic diseases and/or pathological findings present or in history, which might interfere with the drug pharmacokinetics.
* Known history or presence of food allergies or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Acute or chronic diseases and/or clinical finding which may interfere with the aims of the study or with the drug's safety, tolerability, bioavailability and/or pharmacokinetics of the Investigational Medicinal Product (IMP).
* History of kidney disease with impaired renal function.
* History of severe allergy or allergic reactions to the study IMP, its excipients or related drugs, wheat allergy history, allergy to soya and peanut in anamnesis.
* History of unexplained vaginal bleeding.
* Positive result of urine pregnancy test at screening or positive urine pregnancy test at check-in or breastfeeding or lack of results of pregnancy test.
* Benign neoplasms and anamnesis of hyperplastic processes including mastopathy.
* Arterial or venous thromboembolism or thrombophlebitis in anamnesis.
* Reporting drug of abuse at screening & positive results of drug of abuse at check-in in each period.
* Positive result of alcohol breath test at check-in.
* The presence of nicotine or cotinine in urine on screening.
* Serious mental disease and/or inability to cooperate with clinical team.
* Sitting blood pressure after a minimum of 5 minutes of rest is out of the range of 90-140 mmHg for systolic BP and/or 60-90 mmHg for diastolic BP and/or heart rate out of the range of 50-100 bpm during the screening procedure.
* Body temperature is out of the range of 35.7-37.6°C at screening.
* Orthostatic hypotension during screening procedure or in the history.
* Reporting drugs or alcohol (of≥ 40 g per day pure ethanol), solvents or caffeine abuse at screening and check-in in each period.
* Donation of at least 400 ml of blood within 60 days, more than 150 ml of blood within 30 days or more than 100 ml blood plasma or platelets within 14 days before study Period I.
* Following a special diet (e.g. vegetarian) or dieting one month before the study initiation
* Less than 80 days between exit procedure in previous study and the first dosing in this study.
* Any significant clinical abnormality including Hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV), and / or (human immunodeficiency virus) HIV. (On screening)
* Abnormal kidney and/or liver function tests and being assessed as clinically significant by the attending physician.(On Screening).
* Results of laboratory tests( including PT and APTT, TT tests also Erythrocyte sedimentation rate (ESR) and Hormones (FSH, LH, Estradiol, Progesterone and Prolactin hormone (PRL) are outside the normal range and being assessed as clinically significant by the attending physician.
* Uric acid level for women > 6.0 mg/dL on screening.
* Previous liver disease or elevations in serum transaminases alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≥1.0 upper limit of normal (ULN) at the screening (ALT for women up to 63 U/L and AST up to 37 U/L).
* The intake of caffeine, xanthenes, or carbon dioxide CO2-containing beverages within 18 hours of drug administration.
* Consumption of alcohol, grapefruit or grapefruit containing products within 7 days of drug administration
* Ingestion of any supplements like vitamins or herbal products within 7 days prior to the initial dose of the study medication.
* Clinically significant illness within 28 days before the first dosing, including major surgery.
* Exhausting physical exercise in the last 48 hours (e.g. weight lifting) or any recent significant change in dietary or exercise habits.
* Abnormal Vital Signs and being assessed as clinically significant by the attending physician.
* Vomiting or diarrhea on admission.
* Use of organ-toxic drugs or systemic drugs known to substantially alter liver metabolism within 80 days before the first dosing.
* Use of any prescription medication for a period of 14 days before the first dosing.
* Any systemic over-the-counter (OTC) drug treatment and/or vitamins and/or herbal treatment and/or food supplements within 14 days before the first dosing.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Inclusion Criteria:
  - Healthy postmenopausal females. Duration of menopause has to be more than 1 year on the day of informed consent.
Enrollment: 48 (Actual)
Dates: Start 2019-12-13 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Cmax | up to 96 hours post-administration
  Maximum plasma concentration
AUC0-last | up to 96 hours post-administration
  Area under the plasma concentration-time curve from 0 hours to the time of last quantified concentration

SECONDARY OUTCOMES:
Tmax. | up to 96 hours post-administration
  Time point of maximum plasma concentration
AUC0→inf | up to 96 hours post-administration
  Area under the plasma concentration-time curve from 0 hours to infinity
Residual area (%). | up to 96 hours post-administration
  Residual area (%).
λz | up to 96 hours post-administration
  Terminal elimination rate constant
t1/2 | up to 96 hours post-administration
  Half-life of drug elimination during the terminal phase

CONTACTS AND LOCATIONS:
Overall Officials: Vlad Udovytskyi, Study Chair — Joint Stock Company "Farmak"
Locations (1):
- Arab Pharmaceutical Industry Consulting/Pharmaceutical Research Unit, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No